CLINICAL TRIAL: NCT03484585
Title: Single Center, Open-label, Non-randomized, Non-placebo-controlled Study to Investigate the Metabolism, Excretion Pattern, Mass Balance, Safety, Tolerability and Pharmacokinetics After Single Administration of 200 mg [14C]Rogaratinib (Oral Solution) in Healthy Male Subjects
Brief Title: Rogaratinib (BAY1163877) Human Mass Balance Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18084; 2017-002777-19 (EudraCT Number)
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Clinical Trial, Phase I; Pharmacokinetics
Keywords: Mass Balance, metabolism and excretion pattern
MeSH Terms: interventions — Rogaratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rogaratinib (BAY1163877) (Experimental): Healthy male subjects
  Interventions: Drug: Rogaratinib (BAY1163877)

INTERVENTIONS:
Drug: Rogaratinib (BAY1163877) — Single dose, intake orally, 200 mg

SUMMARY:
The objective of this study is to determine the mass balance and routes of excretion of total radioactivity after a single oral 200 mg dose of [14C]rogaratinib given as a solution. For further clinical development, human mass balance data are required to elucidate the absorption, distribution, metabolism, and excretion (ADME) of rogaratinib.

ELIGIBILITY:
Inclusion Criteria:

* The written informed consent must be signed before any study specific tests or procedures are done
* Age: 21 to 65 years (inclusive) at the first screening examination visit
* Body mass index (BMI) 18.5 to 32.0 kg/m2 (both inclusive) and a total body weight of 55 to 100 kg (both inclusive)
* Healthy male subject, as determined by a responsible and experienced physician, based on a medical evaluation including medical history, laboratory tests, physical, cardiac and full ophthalmologic examination
* Subjects of reproductive potential with a partner of child-bearing potential must agree to use adequate contraception when sexually active. This applies from signing of the ICF until 3 months after the study drug administration. The definition of adequate contraception will be based on the judgment of the investigator and on local requirements. Acceptable methods of contraception include, but are not limited to, (i) condoms (male or female, should not be used together) with or without a spermicidal agent; (ii) diaphragm or cervical cap with spermicide; (iii) intra-uterine device; (iv) hormone-based contraception. Subjects must agree to utilize two reliable and acceptable methods of contraception simultaneously. This is not required if safe contraception is achieved by a permanent method, such as vasectomy of the subject or bilateral fallopian tube blockage of the subject's partner; OR if the subject has no requirement for contraception (e.g. same sex partners).
* Ability to understand and follow study-related instructions

Key Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Known or suspected hypersensitivity to rogaratinib or to excipients in the formulation, or to any FGFR inhibitor
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Relevant diseases within the last 4 weeks prior to the first study drug administration
* Current diagnosis of any retinal detachment, retinal pigment epithelial detachment (RPED), serous retinopathy or retinal vein occlusion
* Presence of high myopia or pathological myopia (defined as spherical equivalent ≥ 6.00D), or any retinal abnormalities consistent with pathologic myopia
* Known recent use of recreational drugs (last 3 months), suspicion of drug or alcohol abuse, or positive results of the urine drug or alcohol screen at screening or baseline
* Use of any medication within 14 days before administration of the study drug except paracetamol
* Smoking more than 5 cigarettes daily
* Exposure to radiation for diagnostic reasons (except dental X rays and plain X rays of thorax and bony skeleton [excluding spinal column]), during work or during participation in a clinical study in the period of 1 year prior to screening
* Participation in another study with a radiation burden of > 0.1 mSv and ≤ 1 mSv in the period of 1 year prior to screening; a radiation burden of > 1.1 mSv and ≤ 2 mSv in the period of 2 years prior to screening; a radiation burden of > 2.1 mSv and ≤ 3 mSv in the period of 3 years prior to screening, etc (add 1 year per 1 mSv)
* Previous (within the preceding 3 months; end of previous study to first treatment of the current study) or concomitant participation in another clinical study with investigational medicinal product(s)

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
Cmax of rogaratinib in plasma | At pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 and 168 h post-dose. Collection will be extended depending on the radioactivity recovery.
  Cmax: maximum drug concentration in the measured matrix, directly taken from analytical data
AUC(0-tlast) of rogaratinib in plasma | At pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 and 168 h post-dose. Collection will be extended depending on the radioactivity recovery.
  AUC(0-tlast): area under the measured matrix concentration versus time curve to the last data point above the lower limit of quantitation
AUC of rogaratinib in plasma | At pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 and 168 h post-dose. Collection will be extended depending on the radioactivity recovery.
  AUC: area under the measured matrix concentration versus time curve from the first time point (t=0) extrapolated to infinity
Cmax of total radioactivity in plasma and whole blood | At pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 and 168 h post-dose. Collection will be extended depending on the radioactivity recovery.
AUC(0-tlast) of total radioactivity in plasma and whole blood | At pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 and 168 h post-dose. Collection will be extended depending on the radioactivity recovery.
AUC of total radioactivity in plasma and whole blood | At pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 and 168 h post-dose. Collection will be extended depending on the radioactivity recovery.
AE,ur (%) of rogaratinib and its metabolites | In intervals of 12h from Day -1 till Day 2 and in intervals of 24h afterwards: at pre-dose (-12-0h), 0-12, 12-24, 24-48, 48-72, 72-96,96-120, 120-144 and 144-168 hours post dose. Collection will be extended depending on the radioactivity recovery.
  AE,ur: amount excreted into urine from 0 to infinity
AE,fec (%) of rogaratinib and its metabolites | In intervals of 24h at pre dose (-18-0h), 0-24, 24-48, 48-72, 72-96, 96-120, 120-144 and 144-168 hours post dose. Collection will be extended depending on the radioactivity recovery.
  AE,fec: amount excreted into feces from 0 to infinity
AE,vom (%) of rogaratinib and its metabolites, if applicable | During the first 6 hours after dosing
  AE,vom: amount excreted into vomit

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- PRAHealthSciences, Groningen, Netherlands